CLINICAL TRIAL: NCT00180362
Title: Is Extensive Electrophysiological Testing Before, During and After ICD-Implantation Still Necessary in Patients After Survived Cardiac Arrest? A Prospective Randomised Multi-centre Trial.
Brief Title: Quick ICD Study: Is Extensive Electrophysiological Testing Before, During and After ICD-Implantation Still Necessary ?
Acronym: Quick ICD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Version vom 31.3.1999
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Methods

INTERVENTIONS:
Device: procedure

SUMMARY:
The purpose of this study is to evaluate the strategy of implanting an ICD with or without EPS before, during and after ICD-implantation in a randomised controlled trial, using a combined endpoint of major ICD-related adverse events as the primary outcome measure.

DETAILED DESCRIPTION:
Usually, EPS before and during ICD-implantation is performed to allow risk stratification, to test serial antiarrhythmic drugs, to find suitable ablation sites in patients with hemo-dynamically stable monomorphic VTs, to exclude supraventricular tachycardias as a cause of cardiac arrest and to help programming detection rate and enhancement criteria in the ICD. However, routine EPS preceeding ICD-implantation exposes the patient to some risk and the health care system to considerable costs. So the question has been raised, whether such testing is still necessary and costseffective, if the indiaction for ICD-implantation is clear on a clinical ground.The purpose of this study is to evaluate the strategy of implanting an ICD with or without EPS before during and after ICD-implantation in a randomised controlled trial, using a combined endpoint of major ICD-related adverse events as the primary outcome measure (see details under "Endpoints"). The results will be viewed against the extra costs and patients´ quality of life both study arms.Secondary outcomes are considered as differences in decisions between the groups and difference of events in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* structural heart disease and survived cardiac arrest or hemodynamically unstable VT (bpm > 200/min)

Exclusion Criteria:

* conditions, which make a secondary cause for cardiac arrest probable or are not compatible with a single chamber ICD; co-morbidity, prior ICD PM, or EPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-05; Study Completion 2004-09

PRIMARY OUTCOMES:
Combined endpoint of major ICD-related adverse events as the primary outcome measure

SECONDARY OUTCOMES:
Costs, quality of life, differences in decision making, cardiovascular events , 18 months FU

CONTACTS AND LOCATIONS:
Overall Officials: K. H Kuck, MD, Principal Investigator — Allg. Krankenhaus St. Georg
Locations (1):
- Allg. Krankenhaus St. Georg, Hamburg, Germany